CLINICAL TRIAL: NCT03392805
Title: Infectious Diseases and Movement Program: Study of the Effects of Physical Activity on HIV Infection
Acronym: PRIMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giancarlo Ceccarelli, Reasercher co-PI, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPHID-UniRoma04
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sedentary life style (Experimental)
  Interventions: Behavioral: physical activity
- physically active life style (No Intervention)

INTERVENTIONS:
Behavioral: physical activity — beginning of regular physical activity under the supervision of a coach
  Arms: sedentary life style

SUMMARY:
exercise and physical activity can have an anti-inflammatory effect, while there is evidence that a sedentary lifestyle could be the basis for the development of systemic inflammation and increased cardiovascular risk. The primary objective is to assess whether regular physical activity is able to induce a decrease in systemic immune-activation in HIV positive patients.

DETAILED DESCRIPTION:
Many studies document that exercise and physical activity can have an anti-inflammatory effect, while there is evidence that a sedentary lifestyle could be the basis for the development of systemic inflammation and increased cardiovascular risk. This occurs because a sedentary lifestyle leads to the accumulation of visceral fat, and this is accompanied by an increase in adipokine release and infiltration of adipose tissue by the pro-inflammatory immune cells. Furthermore, the imbalance between immune processes and metabolic processes is associated with the development of insulin resistance, atherosclerosis and neurodegeneration.

The primary objective is to assess whether regular physical activity is able to induce a decrease in systemic immune-activation in HIV positive patients.

To evaluate this hypothesis, the following parameters will be analyzed: evaluation of immune-activation levels, of metabolic parameters, of cardiac function, of immuno-virological set-up, of dietary intake and of physical performance indices in HIV-positive patients with a sedentary lifestyle; these data will be compared with the values measured in the same HIV positive population with a sedentary lifestyle after three months of regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-60 years
2. Patients who have signed informed consent
3. HIV positive patients
4. Patients who have performed a sports medical examination with ECG and are suitable for non-competitive physical activity.

Exclusion Criteria:

1. Anemia, pregnancy or any other contraindication to blood sampling and sports activity
2. Patients suffering from cardiomyopathies and ischemic heart disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Delta between Rockport Walking Test value at T0 and T6 | 6 months

SECONDARY OUTCOMES:
Delta between CD4+CD38+ value at T0 and T6 | 6 months
Delta between CD8+CD38+ value at T0 and T6 | 6 months
Delta between CD4+HLADR+ value at T0 and T6 | 6 months
Delta between CD8+HLADR+ value at T0 and T6 | 6 months
Delta between TNF-α value at T0 and T6 | 6 months
Delta between IL-6 value at T0 and T6 | 6 months
Delta between adiponectin value at T0 and T6 | 6 months
Delta between resistinat T0 and T6 | 6 months
Delta between leptin value at T0 and T6 | 6 months
Delta between maximal Oxygen uptake value at T0 and T6 | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health and Infectious Diseases, University of Rome "La Sapienza", Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided